CLINICAL TRIAL: NCT01091064
Title: IMPACT OF A HEALTH CARE PROTOCOL FOR PATIENTS SUFFERING SYMPTOMS OF MILD ACUTE VIRAL BRONCHIOLITIS ON EARLY DISCHARGE IN THE EMERGENCY DEPARTMENT.
Brief Title: Impact Of A Health Care Protocol For Patients Suffering Symptoms Of Mild Acute Viral Bronchiolitis On Early Release In The Emergency Department
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped because it was not approved for funding
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Dre Chantal Guimont, Professeur, Laval University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 20636
Record Dates: First submitted 2010-03-19; First posted 2010-03-23 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early depart (Experimental): Patients who will be liberated at triage with mild acute viral bronchiolitis
  Interventions: Other: Randomization early depart
- Medical visit group (No Intervention): Patients with acute viral bronchiolitis who will wait to be seen by the physician

INTERVENTIONS:
Other: Randomization early depart — Patients will be randomized to either an early depart or for being seen by a physician.
  Arms: Early depart

SUMMARY:
Acute viral bronchiolitis is the principal cause of lower respiratory tract infection in infants worldwide. It is characterized by a first episode of respiratory distress preceded by rhinorrhea, cough and fever. The majority of patients present with mild symptoms which can be treated safely at home by parents. Every year between October thru April emergency departments in North America are overwhelmed with patients waiting to be seen with mild respiratory infections, such as bronchiolitis. Thus new strategies in health care have to be elaborated to reduce costs and waiting time in the emergency department.

The investigators hypothesize that patients liberated from triage with mild acute viral bronchiolitis would have the same rate of office re-visits than those with mild acute bronchiolitis in the emergency department.

DETAILED DESCRIPTION:
Acute viral bronchiolitis constitutes the principal cause of acute lower respiratory tract infections in infants and children in Nord America. Every year 11% of infants younger than 1 year and 6% of those between 1 and 2 years are affected. Acute viral bronchiolitis is characterized by a first episode of respiratory distress associated to rhinorrhea, cough and fever, other symptoms such as vomiting, use of accessory intercostal muscles and irritability can be present. Mild symptoms presentation in bronchiolitis is very common, these patients do not require treatment or testing, only appropriate information on how to ameliorate respiratory symptoms and a well list of alarm signs for parents are frequently enough to send the patient home.

Increasing workload in the ED is a national worry after the last 20 years. Between October and April, this phenomena is seen each year due to cold and influenza season. From an economic perspective along with a lack in human resources, new strategies have to be implemented to reduce duration and costs in office visits in the emergency department. Since mild bronchiolitis does not require a specific treatment, we hypothesize that patients liberated from triage with mild acute viral bronchiolitis would have the same rate of office re-visits than those with mild acute bronchiolitis in the emergency department.

Our principal objective will be to compare between groups of infants with mild acute viral bronchiolitis the use of hospital resources within the fist 15 days after recruitment. Specific objectives will be to compare between the 2 groups the rate of office re-visit, or to the ED during the fist 15 days after recruitment, the severity of respiratory symptoms during re-visits, on follow up at 2-4 days, 6-8 days and 13-15 days, patient and parent satisfaction of the first visit and of follow up at 2-4 days, 6-8 days and 13-15 days.

This research project will have a rapid and direct effect on quality of health care in infants with acute viral bronchiolitis and their parents, as well as important repercussions on the workload in the waiting rooms of EDs allowing physicians to concentrate on other patients are in need of a rapid attention. This project will be carried on in two high concentration specialized hospitals in the province of Quebec, Canada.

ELIGIBILITY:
Inclusion Criteria:

* patients of any sex aged 3 to 12 months old with the diagnosis of mild acute viral bronchiolitis.

Exclusion Criteria:

* Infants aged < 3 months of > 13 months old.
* Infants born before 30 weeks gestation.
* Infants' weight < 5 kg.
* Infants with a dehydration score of more or equal to 1.
* Yale score > 10.
* Infants with chronic pulmonary, cardiovascular or neuromuscular disease.
* Infants with primary or secondary immunodeficiencies.
* Patients with the antecedent of wheezing.
* Need of any ventilatory support.
* Patients in whom the diagnosis of acute viral bronchiolitis is not precise.
* Patients in whose parents refuse to sign the consent formulary or not willing to participate.

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
emergency revisit rate | 15 days
  emergency revisit rate in the first 15 days after recruitment

CONTACTS AND LOCATIONS:
Locations (1):
- Laval University Hospital Center, Québec, Quebec, Canada